CLINICAL TRIAL: NCT03685682
Title: Safety and Immunogenicity of Non-live, Recombinant Subunit Herpes Zoster Vaccine in VZV-seronegative Solid Organ Transplant Recipients
Brief Title: Recombinant Subunit Herpes Zoster Vaccine in VZV-Seronegative Organ Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Deepali Kumar, Principal Investigator, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UHNTID007
Record Dates: First submitted 2018-09-23; First posted 2018-09-26 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Varicella Zoster Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VZV seronegative Transplant Patients (Experimental): recombinant subunit Herpes zoster vaccine
  Interventions: Biological: recombinant subunit Herpes zoster vaccine

INTERVENTIONS:
Biological: recombinant subunit Herpes zoster vaccine — Seronegative Solid Organ Transplant patients will receive two doses of the subunit Herpes zoster vaccine at 0 and 2-6 months

SUMMARY:
The investigators plan to study the immunogenicity of the vaccine in VZV-seronegative solid organ transplant recipients. VZV-seronegative patients will be enrolled after organ transplantation. The investigators hypothesize that the recombinant subunit Herpes zoster vaccine is able to induce cellular immunogenicity after transplantation in VZV-seronegative patients.

DETAILED DESCRIPTION:
Solid organ transplant recipients receive lifelong immunosuppression and are at increased risk for severe primary VZV infection (chickenpox) and VZV reactivation (shingles). A non-live, recombinant subunit Herpes zoster vaccine (Shingrix; GSK vaccines) was recently licensed for the prevention of shingles in people aged 50 years or older and was shown to induce both cellular and humoral immunity. As both components of the immune system are important for protection against VZV, the investigators plan to study the humoral and cellular immunogenicity of the vaccine after organ transplantation in VZV-seronegative patients. Indeed, the current live VZV vaccine is contraindicated after transplantation; therefore, the non-live recombinant varicella-zoster subunit vaccine, if shown to induce cellular and humoral immunity, could potentially be offered to VZV-seronegative transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Solid organ transplant recipient.
* Age ≥18 years
* VZV-seronegative at time of transplant
* ≥90 days post-transplant
* Able to provide informed consent

Exclusion Criteria:

* Has already received the recombinant subunit Herpes zoster vaccine in the past
* Ongoing CMV viremia > 200 IU/mL
* HIV infection
* Diagnosis of malignancy (e.g. PTLD)
* History of a severe allergic reaction (anaphylactic reaction) after any vaccine
* Documented Chickenpox or Shingles after transplantation
* Congenital immunodeficiency (e.g., CVID)
* Treatment for rejection in the past 30 days
* Immunoglobulin in the past 30 days or anticipated to receive immunoglobulin
* Anti-CD20 monoclonal antibody in the past 6 months or anticipated to receive Anti-CD20 monoclonal antibody
* Plasmapheresis in the past 30 days or anticipated to receive plasmapheresis
* Febrile illness in the past one week
* Unable to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
Humoral immunity to varicella zoster induced by the recombinant subunit Herpes zoster vaccine. | 4 weeks after second dose of vaccine
  Fold increase in concentration of anti-gE antibody titer from pre- to post-vaccination

SECONDARY OUTCOMES:
Rate of Vaccine-related Adverse Events | Up to 4 weeks after second dose of vaccine
  Adverse events will be graded as mild, moderate, severe

CONTACTS AND LOCATIONS:
Overall Officials: Deepali Kumar, MD, Principal Investigator — Multi organ transplant program, University Health Network, Toronto
Locations (1):
- University Health Network, Toronto General Hospital, Multi-Organ Transplant, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] L'Huillier AG, Hirzel C, Ferreira VH, Ierullo M, Ku T, Selzner N, Schiff J, Juvet S, Miao C, Schmid DS, Humar A, Kumar D. Evaluation of Recombinant Herpes Zoster Vaccine for Primary Immunization of Varicella-seronegative Transplant Recipients. Transplantation. 2021 Oct 1;105(10):2316-2323. doi: 10.1097/TP.0000000000003621. PMID 33528118